CLINICAL TRIAL: NCT00275366
Title: Upper Extremity Robotics in Musculoskeletal Rehabilitation
Brief Title: Arm Robotics in Musculoskeletal Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Finley, Margaret - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3827V
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Rotator Cuff Tear
Keywords: cuff, rotator; Rotator cuff
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Device: Robotic Therapy

INTERVENTIONS:
Device: Robotic Therapy

SUMMARY:
This purpose of this study is to determine the outcomes of the first-known application of robotic therapy in the rehabilitation following rotator cuff repair, using a novel vertical oblique robotic module.

DETAILED DESCRIPTION:
Musculoskeletal conditions are a leading cause of disability in the United States accounting for more than 130 million patient visits to healthcare providers annually. Rotator cuff tears are one of the most common causes of pain and disability of the upper extremity. Impaired motor control of the shoulder girdle muscles with concomitant instability often exists prior to any surgical procedure. Re-tears and/or attenuation after rotator cuff repairs occur relatively frequently and may compromise the functional result. Loading of the UE during rehabilitation, thus the repair site, following the surgical procedure has been implicated in these complications Conventional shoulder rehabilitation protocols with the human-human interface do not possess the ability to systematically quantify dosing and progression for patients in the subacute stages thus, potentially overloading the repair site. No evidence-based research exists comparing outcomes of specific rehabilitative training protocols in these post-surgical patients. Consensus statements conclude, �a need for clinical trials, and validated outcome measures is essential�.

Advances in robotics technology offer unprecedented opportunities to improve rehabilitation pathways, but until now these technologies have focused primarily on neurological disease. The MIT Newman Laboratory for Biomechanics and Human Rehabilitation upper extremity (UE) robot is an impedance controlled, back-drivable, oblique-vertical vertical robot that has been designed such that it can safely exert controlled, graded forces to move or guide a limb, functioning in passive, active-assistive, active and resistive modes, providing objective data on the motion. A major advantage is its capacity for real-time, graded changes based on patient input, providing stability against random perturbations, increasing or withdrawing assistance and allowing for dose-specific treatment. The vertical robot device has been shown to be safe and well tolerated without any adverse effects such as shoulder pain.

Goal-directed, quantifiable rehabilitation protocols for redevelopment of function through improved range of motion, strength and motor control are lacking in patients with musculoskeletal impairments. The successful robotic-assisted rehabilitation of the acute and chronic, severe impairment provides an impetus for applying this technology to UE musculoskeletal impairments. The ability to objectively control and measure the dosing and progression during the rehabilitation process is a valuable tool in the advancement of evidence�based rehabilitation interventions The proposed pilot clinical trial will determine if 8-weeks of robotic rehabilitation improves the rate and quality of recovery of range of motion, strength, and function following rotator cuff repair compared with a conventional physical therapy rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

1. aged 40-65 years
2. Surgeon referral with medical clearance;
3. <3 weeks post-arthroscopic rotator cuff repair
4. Rotator cuff tear size <5cm;
5. Surgeon reported good tendon tissue health status
6. Adequate cognition and language skills to provide informed consent and participate in robotics training and/or robotics testing.

Exclusion Criteria:

1. Age <39, or >65 years
2. Rotator cuff tear >5cm
3. Surgical finding of poor tendon tissue status
4. Open surgical procedure;
5. Rotator cuff revision procedure
6. Worker's compensation injury
7. History of neuro-motor disease of the upper extremities.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Finley, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States